CLINICAL TRIAL: NCT02010216
Title: Non-Randomized Phase IV Trial on Efficacy and Safety of Actemra in the Treatment of Adult Patients With Rheumatoid Arthritis
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) in Adult Patients With Rheumatoid Arthritis (SVOBODA Programme)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML23037
Record Dates: First submitted 2013-12-04; First posted 2013-12-12 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- tocilizumab [RoActemra/Actemra] (Experimental): Participants received tocilizumab 8 mg/kg by intravenous infusion every 4 weeks for 12 weeks (3 cycles).
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg by intravenous infusion every 4 weeks
  Other Names: RoActemra/Actemra

SUMMARY:
This open-label, single arm study evaluated the efficacy and safety of RoActemra/Actemra (tocilizumab) in patients with rheumatoid arthritis. Patients received RoActemra/Actemra 8 mg/kg intravenously every 4 weeks, alone or in combination with standard anti-rheumatic therapy, for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥ 18 years of age
* Confirmed moderate or severe rheumatoid arthritis
* Intolerability or absence of effect or decrease in effect of rheumatoid arthritis treatment with disease modifying antirheumatic drugs (DMARDs)

Exclusion Criteria:

* Presence of infectious diseases [tuberculosis (Tb), human immunodeficiency virus (HIV), virus hepatitis A/B/C]
* Inadequate hematologic, renal or liver function
* Peptic ulcer disease (in acute phase)
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Kazakhstan (4):
  - Almaty
  - Astana
  - Shymkent
  - Ust-Kamenogorsk

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tocilizumab [RoActemra/Actemra]
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg by intravenous infusion every 4 weeks for 12 weeks (3 cycles).
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity 28 (DAS28) Score
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
score on a scale | -3.9 (1.1)

2. Primary Outcome: Percentage of Participants Achieving ACR20/50/70 Responses After the Third Infusion Categorized by Highest Response Achieved
Description: American College of Rheumatology (ACR) ACR20, ACR50 or ACR70 response is defined as a ≥ 20% or 50% or 70% improvement (reduction) compared with Baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Baseline, Week 12
Population: Intent-to-treat population included all participants.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
percentage of participants
  ACR20 | 0.0
  ACR50 | 9.5
  ACR70 | 66.7

3. Primary Outcome: Safety: Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events. A SAE was any experience that suggested a significant hazard, contraindication, side effect or precaution that: resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was medically significant.
Time Frame: 12 weeks
Population: Safety population included all participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 23
participants
  AEs | 5
  SAEs | 0

ADVERSE EVENTS:
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 2/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=23)
Drowsiness (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.